CLINICAL TRIAL: NCT04377516
Title: Effects of Specific Pelvic Stabilization Exercise With Transabdominal Ultrasonography-guided Biofeedback in Postpartum Women Suffering From Pregnancy-related Pelvic Girdle Pain
Brief Title: Effects of Specific Pelvic Stabilization Exercise in Postpartum Pregnancy-related Pelvic Girdle Pain Women
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Duplicated with another clinical trial registration.
Sponsor: YI-JU TSAI (Other)
Responsible Party: Sponsor-Investigator, YI-JU TSAI, professor, National Cheng Kung University
Organization: National Cheng Kung University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCKU-TSAI
Record Dates: First submitted 2020-04-28; First posted 2020-05-06 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Pelvic Girdle Pain
MeSH Terms: conditions — Pelvic Girdle Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Transabdominal Sonography-guided Biofeedback group (Experimental): pelvic floor muscle training with transabdominal sonography-guided Biofeedback
  Interventions: Other: pelvic floor muscle training; Other: pelvic floor muscle combined global muscle exercise training; Other: education of pelvic girdle
- Exercise group (Active Comparator): pelvic floor muscle training
  Interventions: Other: pelvic floor muscle training; Other: pelvic floor muscle combined global muscle exercise training; Other: education of pelvic girdle
- Control group (Placebo Comparator): pelvic girdle education
  Interventions: Other: education of pelvic girdle
- Health group (Placebo Comparator): pelvic girdle education
  Interventions: Other: education of pelvic girdle

INTERVENTIONS:
Other: pelvic floor muscle training — pelvic floor muscle training
  Arms: Exercise group; Transabdominal Sonography-guided Biofeedback group
Other: pelvic floor muscle combined global muscle exercise training — pelvic floor muscle combined global muscle exercise training
  Arms: Exercise group; Transabdominal Sonography-guided Biofeedback group
Other: education of pelvic girdle — education of pelvic girdle

SUMMARY:
Postpartum women with PPGP receiving specific pelvic stabilization exercise training with transabdominal sonography-guided Biofeedback would have better improvements on muscle functions, physical functions, pain, and disability compared to the regular pelvic stabilization exercise group

ELIGIBILITY:
Inclusion Criteria:

* postpartum : ≥ 3 months
* pregnancy-related pelvic pain
* pain location is located between posterior iliac crest and gluteal fold
* Clinical screening test for pelvic pain :

ASLR : positive and SI joint ≥ 2 (+ symphysis ≥ 1)

Exclusion Criteria:

* lumbar or pelvic surgery
* other causes of pelvic pain (such as fractures)
* Radiculopathy
* other health problems, such as cancer, cardiovascular disease, rheumatism , etc
* daily activities limited , unable to complete the experiment
* communication disorders
* mental disorder
* pregnancy
* have been trained in stable muscle strength in the past.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Muscle function measures of abdominal muscle | 8 weeks
  Untrasonography image for muscle thickness of abdominal muscle during rest and ASLR test.
Muscle function measures of inter recti distance | 8 weeks
  Untrasonography image for muscle thickness of inter recti distance during rest, maximum contraction, and ASLR test.
Muscle function measures of pelvic floor muscle control | 8 weeks
  Untrasonography image for muscle thickness of pelvic floor muscle control during rest, maximum contraction, and ASLR test.
pain intensity measure of Numeric Rating Scale (NRS) | 8 weeks
  Numeric Rating Scale (NRS) is a self-reported instrument assessing average pain intensity in currently. Possible score range from 0 (no pain) to 10 (worst possible pain).
pain intensity measure of pelvic girdle questionnaire (PGQ) | 8 weeks
  pelvic girdle questionnaire(PGQ) is a self-reported instrument assessing pelvic girdle pain intensity in currently. Questionnaire consisting of 20 activity items and 5 symptom items on a 4-point response scale. Possible score range from 0 (no pain) to 100 (worst possible pain).
pain intensity measure of Oswestry Low Back Pain Disability Questionnaire (ODI) | 8 weeks
  Oswestry Low Back Pain Disability Questionnaire(ODI) is a self-reported instrument assessing patient's permanent functional disability in currently. For each section the total possible score is 5: if the first statement is marked the section score = 0; if the last statement is marked, it = 5. The higher the score, the greater the degree of disability.
functional performance of ASLR fatigue task | 8 weeks
  Participants lifted the heel of the test leg to 20 cm for as long as possible. Participants were required to maintain pressure in the cuff beneath their back as close to 40 mm Hg as possible. Visual feedback of cuff pressure was provided throughout the task, but no instruction was given on how to affect cuff pressure. Task failure was defi ned as an inability to maintain heel height 10 cm or more off the plinth and/or a change in cuff pressure of 20 mm Hg or more.
functional performance of timed up and go test | 8 weeks
  Test instructions were given in Norwegian. Translated into English, the instructions were as follows: 'After "ready, set, go" stand up, walk as fast as you can until you cross the white line, turn around, and walk back to the chair and sit down again'. The white line was positioned 3m from the patient's starting position.
  'After "ready, set, go" stand up, walk as fast as you can until you cross the white line, turn around, and walk back to the chair and sit down again'. The white line was positioned 3m from the patient's starting position.
functional performance of 6m timed walk test(fast walking) | 8 weeks
  Subjects commenced the test in standing with their toes up against the tape marker. Test instructions translated into English were as follows: 'After "ready, set, go", walk as fast as you can up to the last white line without stopping or speaking along the way'. Performances were timed (to the nearest 100th of a second) between the 2m and 8m markers and later converted into speed in metres per second.

SECONDARY OUTCOMES:
General health | 8 weeks
  36-item Short-Form Survey(SF-36)

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University, Tainan, Taiwan